CLINICAL TRIAL: NCT02795182
Title: A Phase 1b, Open Label, Multiple Dose, Dose Escalation and Expansion Study to Assess Safety, Tolerability and Antitumor Activities of the Combination of BGB-3111 With BGB-A317 in Subjects With B-Cell Lymphoid Malignancies
Brief Title: Zanubrutinib (BGB-3111) in Combination With Tislelizumab (BGB-A317) in Participants With B-cell Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111_BGB-A317_Study_001
Record Dates: First submitted 2016-06-04; First posted 2016-06-10 (Estimated); Results first posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-03

CONDITIONS: Lymphoma; Leukemia
Keywords: Relapsed; Refractory
MeSH Terms: conditions — Lymphoma; Leukemia; Recurrence | interventions — zanubrutinib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib abd Tislelizumab (Other): Based on results of the dose escalation cohorts and the identified recommended Phase 2 dose, all patients will receive zanubrutinib at 160 mg orally twice daily in combination with intravenous infusion of tislelizumab 200mg given every 21 days, to be continued until disease progression, unacceptable toxicity, treatment consent withdrawal, or study termination
  Interventions: Drug: Zanubrutinib; Drug: Tislelizumab

INTERVENTIONS:
Drug: Zanubrutinib
  Other Names: BGB-3111; Brukinsa
Drug: Tislelizumab
  Other Names: BGB-A317

SUMMARY:
This study is evaluating the safety and preliminary efficacy of BGB-3111 in combination with BGB-A317 in participants with B-cell lymphoid malignancies.

ELIGIBILITY:
Key Inclusion Criteria

Participants may be entered in the study only if they meet all of the following criteria:

1. Dose escalation for Dose Levels 1, 2, and 3: participants with relapsed or refractory World Health Organization (WHO) classification-defined B-lymphoid malignancy following at least 1 line of therapy, with no therapy of higher priority available, including chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL), mantle cell lymphoma (MCL), follicular lymphoma (FL), human cultured lymphoblast (HCL), Marginal zone lymphoma (MZL), non-germinal center B-cell (GCB) DLBCL, GCB DLBCL, transformed FL, and Richter's transformation (NOTE: participants with WM are excluded from enrollment as of Amendment 3).
2. Dose expansion for Cohorts 1 to 4: participants with either of the following relapsed or refractory WHO-classified lymphoid malignancies who have received at least 1 prior line of standard therapy: a. Cohort 1: GCB DLBCL, with cell of origin defined by either immunohistochemistry or gene expression profiling. b. Cohort 2: non-GCB DLBCL, with cell of origin defined by either immunohistochemistry or gene expression profiling. participants who have transformed to DLBCL from another histology may be enrolled into Cohort 3. c. Cohort 3: Transformed lymphoid malignancy, including but not limited to: i. Large cell transformation of chronic lymphocytic leukemia (Richter's transformation). ii. Large cell transformation of other WHO-classified indolent non-Hodgkin's lymphoma, including FL, or MZL. d. Cohort 4: Histologically confirmed primary central nervous system lymphoma (PCNSL) or secondary central nervous system lymphoma (SCNSL) of breast or testicular origin: i. Must be able to tolerate lumbar puncture and/or Ommaya taps. ii. Must have received at least 1 prior central nervous system (CNS)-directed therapy. iii. Presence of brain parenchymal and/or leptomeningeal disease.
3. Aged ≥ 18 years, able and willing to provide written informed consent and to comply with the study protocol.
4. Measurable disease for non-Hodgkin lymphoma defined as ≥ 1 nodal lesion that is > 15 mm in the longest diameter and can be accurately measured in at least 2 dimensions with computed tomography (CT) scan, or ≥ 1 extra-nodal lesion that is > 10 mm in the longest diameter and can be accurately measured in at least 2 dimensions with CT scan, except for PCNSL or SCNSL.
5. Participants with an accessible tumor lesion must agree to a tumor biopsy at screening and another before the drug administration on Cycle 1 Day 8, ideally taken from the same tumor lesion, for biomarker analysis (up to first 12 qualified participants), except for PCNSL. Additionally, participants with DLBCL must have archival tumor tissue or agree to a tumor biopsy for confirmation of the DLBCL subtype.
6. Laboratory parameters as specified below: a. Hematologic: Platelet count ≥ 50 × 109/L; absolute neutrophil count ≥ 1.0 × 109 cells/L; participants with neutrophils < 1.0 × 109/L unless cytopenias are a direct result of active leukemia or lymphoma, in which case platelet count ≥ 35 × 109/L, absolute neutrophil count ≥ 0.75 × 109/L are allowed. (Note: Platelet transfusion administered ≤ 7 days of screening to raise pre-treatment platelet count to ≥ 35 x 109/L is prohibited.) b. Hepatic: Total bilirubin ≤ 1.5 the upper limit of normal (ULN) or ≤ 2.0 × ULN for participants with Gilbert syndrome, aspartate transaminase (AST), and alanine aminotransaminase (ALT) ≤ 3 × ULN. c. Renal: Creatinine clearance ≥ 30 mL/min (as estimated by the Cockcroft-Gault equation or as measured by nuclear medicine scan or 24-hour urine collection). participants requiring hemodialysis will be excluded.
7. Anticipated survival of at least 4 months.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
9. Female participants of childbearing potential and nonsterile males must practice at least 1 of the following methods of birth control with partner(s) throughout the study and for ≥ 3 months after discontinuing study drug: total abstinence from sexual intercourse, double-barrier contraception, intrauterine device or hormonal contraceptive initiated at least 3 months prior to first dose of study drug.
10. Male participants must not donate sperm from initial study drug administration until 180 days after drug discontinuation.

Key Exclusion Criteria

Participants will not be entered in the study for any of the following reasons:

1. Known, active, CNS lymphoma or leukemia, except for Cohorts 4.
2. Diagnosis with Waldenstrom's macroglobulinemia (WM).
3. For PCNSL and SCNSL (Cohorts 4): a. Require corticosteroid therapy > 16 mg dexamethasone daily or equivalent. b. Corticosteroid therapy ≤ 16 mg dexamethasone daily or equivalent at study entry from which, in the Investigator's opinion, it is expected that the participant cannot be tapered off after the first 4 weeks of study treatment. c. Intraocular PCNSL without evidence of brain disease. d. SCNSL actively receiving treatment for extra-CNS disease. e. PCNSL actively receiving concomitant local or systemic therapy for CNS disease.
4. Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenia purpura.
5. History of stroke or cerebral hemorrhage within 6 months of enrollment.
6. History of significant cardiovascular disease, defined as: a. Congestive heart failure greater than New York Heart Association (NYHA) class II according to the NYHA functional classification. b. Unstable angina or myocardial infarction with 6 months of enrollment. c. Serious cardiac arrhythmia or clinically significant ECG abnormality: corrected QT wave (QTcF) > 480 msec based on the Fridericia's formula or other ECG abnormalities including second-degree atrioventricular block type II, third-degree atrioventricular block. Participants who have a pacemaker will be allowed on study despite ECG abnormalities or the inability to calculate the QTc.
7. Severe or debilitating pulmonary disease (dyspnea at rest, significant shortness of breath, congestive obstructive pulmonary disease).
8. History of severe allergic or anaphylactic reactions to monoclonal antibody therapy.
9. Prior Bruton's tyrosine kinase (BTK) inhibitor or anti-PD-1/anti-PD-L1 treatment.
10. Any illness or condition that in the opinion of the investigator may affect safety of treatment or evaluation of any study endpoint.
11. Active autoimmune diseases or history of severe autoimmune diseases; these include but are not limited to a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis systemic lupus erythematosus, rheumatoid arthritis, connective tissue diseases, scleroderma, inflammatory bowel disease, Crohn's disease, ulcerative colitis, autoimmune hepatitis, toxic epidermal necrolysis, Stevens-Johnson syndrome, or clinically manifest antiphospholipid syndrome. Note: Participants are permitted to enroll if they have vitiligo, eczema, type I diabetes mellitus, or endocrine deficiencies, including thyroiditis managed with replacement hormones including physiologic doses of corticosteroids. Participants with Sjögren's syndrome and psoriasis controlled with topical medication and participants with positive serology, such as antinuclear antibodies or antithyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible.
12. A condition requiring systemic treatment with either corticosteroids (> 20 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of study drug administration, except for PCNSL and SCNSL. Note: adrenal replacement doses ≤ 20 mg daily prednisone or equivalents are permitted in the absence of active autoimmune disease; Participants are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption).
13. History of interstitial lung disease or noninfectious pneumonitis, except for those induced by radiation therapy.
14. Requirement for medications which strong cytochrome P450 (CYP)3A inhibitors or inducers.
15. Vaccination with a live vaccine within 28 days of the initiation of treatment.
16. A candidate for hematopoietic stem cell transplantation. Participants are excluded if they had received an allogeneic stem cell transplantation within 6 months or have active graft-versus-host-disease requiring ongoing immunosuppression.
17. Participated in any investigational drug study within 28 days or not recovered from toxicity of any prior chemotherapy to Grade ≤ 1.
18. History of other active malignancies within 2 years of study entry, with the exception of adequately treated in-situ carcinoma of cervix; localized basal cell or squamous cell carcinoma of skin; or previous malignancy confined and treated locally (surgery or other modality) with curative intent.
19. Major surgery in the past 4 weeks prior to the first day of screening.
20. Active and symptomatic fungal, bacterial, and/or viral infection; human T-cell lymphotropic virus type 1 seropositive status.
21. Human immunodeficiency virus (HIV) infection, or active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] detected. • Hepatitis B/C serologic markers and viral load will be tested at screening. The hepatitis B testing includes HBsAg, HBcAb, and HBsAb as well as hepatitis B virus (HBV) DNA by Polymerase chain reaction (PCR) if the participant is negative for HBsAg but HBcAb positive (regardless of HBsAb status). The hepatitis C testing includes Hepatitis C virus (HCV) antibody as well as HCV RNA by PCR if the Participant is HCV antibody positive. Participants with positive HBsAg and/or detectable level of HBV DNA or detectable level of HCV RNA (≥ 15 IU/mL) are not eligible. Participants negative for HBsAg, HBcAb positive, and HBV DNA negative must undergo monthly HBV DNA screening by PCR. Participants positive for HCV antibody but negative for HCV RNA (defined as < 15 IU) must undergo monthly HCV RNA screening.
22. Inability to comply with study procedures.
23. Pregnant or nursing women.
24. Men or women of childbearing potential who refuse to use an adequate measure of contraception, unless they have past medical history of surgical sterilization.
25. Currently taking or plan to take CNS penetrant therapy such as thiotepa, cytarabine, or partially CNS penetrant agents known to be active in lymphoid tumors, such as rituximab.
26. Has taken or plans to take any chemotherapy, immunotherapy (eg, interleukin, interferon, thymoxin), or any investigational therapies to treat leukemia or lymphoma within 28 days or 5 half-lives (whichever is shorter) of the first study drug administration, including CNS penetrating agents.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — BeiGene
Locations (10):
- Australia (7):
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Concord Hospital, Sydney, New South Wales
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Hospital, Clayton, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Epworth Healthcare, Richmond, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- China (3):
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Shanghai jiaotong university school of medicine Ruijin Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Othman J, Verner E, Tam CS, Huang J, Lin L, Hilger J, Trotman J, Gasiorowski R. Severe hemolysis and transfusion reactions after treatment with BGB-3111 and PD-1 antibody for Waldenstrom macroglobulinemia. Haematologica. 2018 May;103(5):e223-e225. doi: 10.3324/haematol.2017.186817. Epub 2018 Feb 8. No abstract available. PMID 29439186

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of a dose escalation phase during which 3 dose levels of tislelizumab were administered in combination with a total of 320 mg zanubrutinib to determine the recommended phase 2 dose (RP2D). Once RP2D was determined all participants remaining in the study were switched to RP2D. A total of 75 participants were enrolled in both phases combined. As pre-specified in the protocol, analyses were conducted by disease subtype on the overall enrolled participants and not by phases.
Groups:
- Dose Escalation: Zanubrutinib 320 mg QD + Tislelizumab 2.0 mg/kg Q3W: Zanubrutinib 320 mg once daily (QD) orally with tislelizumab 2.0 milligrams/kilogram (mg/kg) intravenously (IV) once every 3 weeks until unresolved toxicity, unacceptable adverse events (AEs) or discontinuation by sponsor.
- Dose Escalation: Zanubrutinib 320 mg QD + Tislelizumab 5.0 mg/kg Q3W: Zanubrutinib 320 mg QD orally with tislelizumab 5.0 mg/kg IV once every 3 weeks until unresolved toxicity, unacceptable AEs or discontinuation by sponsor.
- Dose Escalation: Zanubrutinib 160 mg BID + Tislelizumab 200 mg Flat Q3W: Zanubrutinib 160 mg twice daily (BID) orally with tislelizumab 200 mg flat dose IV once every 3 weeks until unresolved toxicity, unacceptable AEs or discontinuation by sponsor
- Dose Expansion: Zanubrutinib 160 mg BID + Tislelizumab 200 mg Flat Q3W: Zanubrutinib 160 mg BID orally with tislelizumab 200 mg flat dose IV once every 3 weeks until unresolved toxicity, unacceptable AEs or discontinuation by sponsor
Period: Overall Study
Arm/Group | Dose Escalation: Zanubrutinib 320 mg QD + Tislelizumab 2.0 mg/kg Q3W | Dose Escalation: Zanubrutinib 320 mg QD + Tislelizumab 5.0 mg/kg Q3W | Dose Escalation: Zanubrutinib 160 mg BID + Tislelizumab 200 mg Flat Q3W | Dose Expansion: Zanubrutinib 160 mg BID + Tislelizumab 200 mg Flat Q3W
Started | 15 | 10 | 7 | 43
Completed | 0 | 0 | 0 | 0
Not Completed | 15 | 10 | 7 | 43
Not completed — Death | 5 | 4 | 4 | 18
Not completed — Sponsor's Decision at Discontinuation and Death at End of Trial | 0 | 0 | 0 | 1
Not completed — Physician's decision at Discontinuation and Death at End of Trial | 0 | 0 | 0 | 2
Not completed — Study Ended by Sponsor Once Primary and Secondary Objectives Were Met | 3 | 2 | 0 | 8
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Roll Over to Long Term Extension | 3 | 3 | 2 | 5
Not completed — Progressive Disease | 0 | 1 | 0 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set includes all participants who receive at least 1 dose of zanubrutinib and/or tislelizumab.
Groups:
- Dose Escalation: Zanubrutinib 320 mg QD + Tislelizumab 2.0 mg/kg Q3W: Zanubrutinib 320 mg QD orally with tislelizumab 2.0 mg/kg IV once every 3 weeks until unresolved toxicity, unacceptable AEs or discontinuation by sponsor.
- Dose Escalation: Zanubrutinib 160 mg BID + Tislelizumab 200 mg Flat Q3W; Dose Expansion: Zanubrutinib 160 mg BID + Tislelizumab 200 mg Flat Q3W: Zanubrutinib 160 mg BID orally with tislelizumab 200 mg flat dose IV once every 3 weeks until unresolved toxicity, unacceptable AEs or discontinuation by sponsor
- Total: Total of all reporting groups
Arm/Group | Dose Escalation: Zanubrutinib 320 mg QD + Tislelizumab 2.0 mg/kg Q3W | Dose Escalation: Zanubrutinib 320 mg QD + Tislelizumab 5.0 mg/kg Q3W | Dose Escalation: Zanubrutinib 160 mg BID + Tislelizumab 200 mg Flat Q3W | Dose Expansion: Zanubrutinib 160 mg BID + Tislelizumab 200 mg Flat Q3W | Total
Number analyzed (Participants) | 15 | 10 | 7 | 43 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (12.63) | 60.7 (6.52) | 70.4 (5.26) | 66.7 (9.85) | 65.0 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 4 | 16 | 29
  Male | 11 | 5 | 3 | 27 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 12 | 7 | 7 | 38 | 64
  Unknown or Not Reported | 3 | 3 | 0 | 4 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race- White | 14 | 9 | 7 | 33 | 63
  Race - Asian | 1 | 1 | 0 | 9 | 11
  Race - Other | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation: Maximum Tolerated Dose (MTD) of Tislelizumab
Description: The MTD of tislelizumab is considered the dose level below that at which at least 2 participants (or at least 33%) experience a dose-limiting toxicity (DLT).
Time Frame: From the date of first dose of study drugs until RP2D was determined (Approximately 1 year and 10 months)
Population: Dose Escalation Phase: Safety analysis set: Includes all participants who receive at least 1 dose of zanubrutinib and/or tislelizumab.
Measure: Number; unit: mg
Groups:
- Dose Escalation Phase: Participants received either zanubrutinib 320 mg once daily orally in combination with tislelizumab 2.0 mg/kg IV once every 3 weeks, or zanubrutinib 320 mg once daily orally with tislelizumab 5.0 mg/kg IV once every 3 weeks or zanubrutinib 160 mg twice daily orally with tislelizumab 200 mg flat dose IV once every 3 weeks unresolved toxicity, unacceptable adverse events (AEs) or discontinuation by sponsor
Arm/Group | Dose Escalation Phase
Number analyzed (Participants) | 32
mg | NA — MTD not reached because number of participants with dose limiting toxicities (DLTs) per dose level did not reach the required threshold.

2. Primary Outcome: Dose Escalation: RP2D of Tislelizumab
Description: The RP2D of tislelizumab in combination with zanubrutinib will be selected by taking into account the safety, tolerability, and pharmacokinetic (PK) profile.
Time Frame: From the date of first dose of study drugs until final R2PD was decided (Approximately 1 year and 10 months)
Population: Dose Escalation Phase: Safety analysis set: Included all participants who receive at least 1 dose of zanubrutinib and/or tislelizumab.
Measure: Number; unit: mg
Arm/Group | Dose Escalation Phase
Number analyzed (Participants) | 32
mg | 200

3. Secondary Outcome: Number of Participants With TEAEs and SAEs
Description: A treatment-emergent adverse event (TEAE) was defined as an AE that had an onset date during the treatment emergent period, defined as from the first dose date of zanubrutinib or tislelizumab (whichever is earlier) through 30 days after the last dose (permanent discontinuation of study drug) of zanubrutinib or 90 days after the last dose of tislelizumab, whichever is later, or prior to initiation of new anti-cancer therapy. Treatment-related serious adverse events (SAEs) and any worsening of a TEAE by PT post treatment-emergent period were also counted as TEAEs.
Time Frame: From the day of first dose of study drug until end of study (up to 4 years and 6 months)
Population: Safety Analysis Set
Measure: Number; unit: Number of participants
Arm/Group | Dose Escalation: Zanubrutinib 320 mg QD + Tislelizumab 2.0 mg/kg Q3W | Dose Escalation: Zanubrutinib 320 mg QD + Tislelizumab 5.0 mg/kg Q3W | Dose Escalation: Zanubrutinib 160 mg BID + Tislelizumab 200 mg Flat Q3W | Dose Expansion: Zanubrutinib 160 mg BID + Tislelizumab 200 mg Flat Q3W
Number analyzed (Participants) | 15 | 10 | 7 | 43
Number of participants
  Participants With at Least One TEAE | 15 | 9 | 7 | 40
  Participants With at Least One SAE | 10 | 10 | 4 | 23

4. Secondary Outcome: Overall Response Rate
Description: ORR, is defined as the percentage of participants who had complete response (CR) or partial response (PR) by standard disease-specific response criteria. for WM participants ORR includes minor response (MR) and very good partial response (VGPR).
Time Frame: Up to 4 years and 6 months
Population: Safety analysis set : Includes all participants who receive at least 1 dose of zanubrutinib and/or tislelizumab. Per protocol Safety analysis set was used for all safety and efficacy outcome analyses. All efficacy analyses were done by disease type for both part 1 and part 2 combined and not by dose level as specified in the protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Other B-Cell Malignancies: Zanubrutinib 160 mg twice daily orally with tislelizumab 200 mg flat dose IV once every 3 weeks until unresolved toxicity, unacceptable AEs or discontinuation by sponsor. This group included participants with CLL/SLL, WM, FL, MCL and MZL.
- GCB DLBCL; Non-GCB DLBCL; Richter's Transformation; Transformed Lymphoid Malignancy; PCNSL or SCNSL of Breast or Testicular Origin: Zanubrutinib 160 mg twice daily orally with tislelizumab 200 mg flat dose IV once every 3 weeks until unresolved toxicity, unacceptable AEs or discontinuation by sponsor
Arm/Group | Other B-Cell Malignancies | GCB DLBCL | Non-GCB DLBCL | Richter's Transformation | Transformed Lymphoid Malignancy | PCNSL or SCNSL of Breast or Testicular Origin
Number analyzed (Participants) | 16 | 12 | 15 | 7 | 20 | 5
Percentage of participants | 37.5 [15.2 to 64.6] | 25.0 [5.5 to 57.2] | 40.0 [16.3 to 67.7] | 42.9 [9.9 to 81.6] | 40 [19.1 to 63.9] | 40 [5.3 to 85.3]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the date that a confirmed objective response is first documented to the date of progressive disease (PD) or death due to any cause for those participants with a confirmed PR or CR.
Time Frame: Up to 4 years and 6 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Other B-Cell Malignancies | GCB DLBCL | Non-GCB DLBCL | Richter's Transformation | Transformed Lymphoid Malignancy | PCNSL or SCNSL of Breast or Testicular Origin
Number analyzed (Participants) | 16 | 12 | 15 | 7 | 20 | 5
Months | 22.36 [7.72 to NA] — NA = Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA = Not estimable due to insufficient number of participants with events | 6.79 [2.36 to NA] — NA = Not estimable due to insufficient number of participants with events | 17.47 [2.96 to NA] — NA = Not estimable due to insufficient number of participants with events | 8.89 [2.83 to NA] — NA = Not estimable due to insufficient number of participants with events | 7.80 [7.06 to 8.55]

6. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS, is defined as the time from the first dose of study medication to objective disease progression or death
Time Frame: Up to 4 years and 6 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Other B-Cell Malignancies | GCB DLBCL | Non-GCB DLBCL | Richter's Transformation | Transformed Lymphoid Malignancy | PCNSL or SCNSL of Breast or Testicular Origin
Number analyzed (Participants) | 16 | 12 | 15 | 7 | 20 | 5
Months | 16.94 [5.39 to NA] — NA = Not estimable due to insufficient number of participants with events | 1.43 [0.57 to NA] — NA = Not estimable due to insufficient number of participants with events | 2.80 [1.43 to 6.99] | 2.93 [2.43 to 20.33] | 4.68 [1.26 to 8.52] | 8.42 [0.33 to 16.07]

7. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) to Tislelizumab
Time Frame: From the day of first dose of study drug until end of study (up to 4 years and 6 months)
Population: Safety analysis set included all participants who received at least 1 dose of tislelizumab. N is the number of evaluable participants. Evaluable participants received at least one complete dose of Tislelizumab and for whom one baseline ADA and at least one post dose ADA values are available.
Measure: Number; unit: Number of participants
Arm/Group | Dose Escalation: Zanubrutinib 320 mg QD + Tislelizumab 2.0 mg/kg Q3W | Dose Escalation: Zanubrutinib 320 mg QD + Tislelizumab 5.0 mg/kg Q3W | Dose Escalation: Zanubrutinib 160 mg BID + Tislelizumab 200 mg Flat Q3W | Dose Expansion: Zanubrutinib 160 mg BID + Tislelizumab 200 mg Flat Q3W
Number analyzed (Participants) | 3 | 4 | 5 | 35
Number of participants
  Treatment Emergent ADA | 0 | 0 | 0 | 1
  Neutralizing antibody Positive | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the Day of first dose of study drug until end of Study (up to 4 years and 6 months)
Description: Safety analysis set: Includes all participants who receive at least 1 dose of zanubrutinib and/or tislelizumab
Groups:
- Dose Escalation: Zanubrutinib 320 mg QD + Tislelizumab 2.0 mg/kg: Zanubrutinib 320 mg QD orally with tislelizumab 2.0 mg/kg IV once every 3 weeks until unresolved toxicity, unacceptable AEs or discontinuation by sponsor.
- Dose Escalation: Zanubrutinib 320 mg QD + Tislelizumab 5.0 mg/kg: Zanubrutinib 320 mg QD orally with tislelizumab 5.0 mg/kg IV once every 3 weeks until unresolved toxicity, unacceptable AEs or discontinuation by sponsor.
Arm/Group | Dose Escalation: Zanubrutinib 320 mg QD + Tislelizumab 2.0 mg/kg | Dose Escalation: Zanubrutinib 320 mg QD + Tislelizumab 5.0 mg/kg | Dose Escalation: Zanubrutinib 160 mg BID + Tislelizumab 200 mg Flat Q3W | Dose Expansion: Zanubrutinib 160 mg BID + Tislelizumab 200 mg Flat Q3W
All-Cause Mortality (participants affected / at risk) | 5/15 | 4/10 | 4/7 | 21/43
Serious Adverse Events (participants affected / at risk) | 10/15 | 10/10 | 4/7 | 23/43
Other Adverse Events (participants affected / at risk) | 15/15 | 9/10 | 7/7 | 40/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation: Zanubrutinib 320 mg QD + Tislelizumab 2.0 mg/kg (N=15) | Dose Escalation: Zanubrutinib 320 mg QD + Tislelizumab 5.0 mg/kg (N=10) | Dose Escalation: Zanubrutinib 160 mg BID + Tislelizumab 200 mg Flat Q3W (N=7) | Dose Expansion: Zanubrutinib 160 mg BID + Tislelizumab 200 mg Flat Q3W (N=43)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atypical haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymph gland infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Urinary tract infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Viral rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemolytic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autonomic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalitis autoimmune (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation: Zanubrutinib 320 mg QD + Tislelizumab 2.0 mg/kg (N=15) | Dose Escalation: Zanubrutinib 320 mg QD + Tislelizumab 5.0 mg/kg (N=10) | Dose Escalation: Zanubrutinib 160 mg BID + Tislelizumab 200 mg Flat Q3W (N=7) | Dose Expansion: Zanubrutinib 160 mg BID + Tislelizumab 200 mg Flat Q3W (N=43)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 9 (21)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (33)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 1 (2) | 0 (0) | 9 (21)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (5) | 0 (0) | 7 (10)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Coeliac disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 9 (10)
Diarrhoea (Gastrointestinal disorders) | 6 (10) | 2 (2) | 2 (2) | 10 (14)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Lip ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 1 (1) | 7 (9)
Oral blood blister (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue geographic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 8 (12)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (5) | 2 (2) | 0 (0) | 9 (12)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site irritation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Pyrexia (General disorders) | 3 (3) | 1 (2) | 0 (0) | 3 (4)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Campylobacter sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ludwig angina (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail bed infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 3 (3) | 1 (1) | 5 (7)
Urinary tract infection (Infections and infestations) | 1 (7) | 0 (0) | 2 (3) | 6 (18)
Viral rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Vulvitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (5) | 0 (0) | 10 (14)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Human metapneumovirus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (13)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 3 (27)
Platelet count decreased (Investigations) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Serum ferritin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 1 (1) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 6 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0) | 3 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 4 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 5 (8)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (6)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (6)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 4 (5)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 0 (0) | 7 (10)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (3) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (5) | 1 (2) | 2 (3) | 3 (5)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 3 (3)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT02795182/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT02795182/SAP_001.pdf